CLINICAL TRIAL: NCT02959749
Title: Phase III Study of Osimertinib or Docetaxel-bevacizumab as Third-line Treatment in EGFR T790M Mutated Non-Small Cell Lung Cancer
Brief Title: Osimertinib or Docetaxel-bevacizumab as Third-line Treatment in EGFR T790M Mutated Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, Director, Qingdao Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QingdaoCH20161101
Record Dates: First submitted 2016-11-05; First posted 2016-11-09 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2016-11

CONDITIONS: Progression Free Survival
Keywords: Osimertinib; EGFR T790M Resistant Mutation; Docetaxel; Bevacizumab; Non Small Cell Lung
MeSH Terms: interventions — osimertinib; Docetaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel, bevacizumab (Active Comparator): docetaxel, 75mg/m2, intravenous infusion on day 1. VEGF monoclonal antibody bevacizumab, 7.5 mg/m2, intravenous infusion on day 1, every 21days a cycle，until disease progression, intolerable toxicities, or patient death.
  Interventions: Drug: docetaxel, bevacizumab
- EGFR TKI (Experimental): osimertinib 80mg oral once daily，until disease progression, intolerable toxicities, or patient death.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — 80 mg oral daily; until disease progression, intolerable toxicities, or patient death.
  Arms: EGFR TKI
Drug: docetaxel, bevacizumab — Docetaxel and bevacizumab are common used in third line therapy in non-small cell lung cancer if not used before. Docetaxel (75 mg/m2) intravenous infusion on day 1 and bevacizumab (7.5 mg/kg) on day 1 every 21days a cycle, until disease progression, intolerable toxicities, or patient death.
  Arms: Docetaxel, bevacizumab

SUMMARY:
Acquired epidermal growth factor receptor (EGFR) T790M mutation is the most common genetic change after resistant to first generation EGFR tyrosine kinase inhibitor (EGFR TKI) in non-small cell lung cancer. After a 10 to 14 months median progression-free survival with the treatment of first generation EGFR TKI, half of patients will get disease progression.For patients progression after treated with first line EGFR TKI and second line double bullets chemotherapy or chemotherapy then EGFR TKI, optimal third line therapy is quite critical important for benefit patients' survival. We conducted this study was aimed to compare the efficacy and toxicity between osimertinib and docetaxel-bevacizumab as the third line therapy in patients with local advanced or metastatic non-squamous cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* local advanced or metastatic non-small cell lung cancer
* large cell lung carcinoma or adenocinoma
* Previously treated by TKI-Chemotherapy or Chemotherapy-TKI
* EGFR T790M positive
* No uncontrolled hypertension
* No active bleeding or thrombosis in recent 6 months
* No previously treated with VEGF antibody

Exclusion Criteria:

* newly diagnosed thrombosis
* anti-coagulation therapy
* uncontrolled hypertension
* uncontrolled nephropathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-08; Primary Completion 2017-10 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
progression free survival | Average 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao Central Hospital, Qingdao Cancer Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nie K, Zhang Z, Zhang C, Geng C, Zhang L, Xu X, Liu S, Wang S, Zhuang X, Lan K, Ji Y. Osimertinib compared docetaxel-bevacizumab as third-line treatment in EGFR T790M mutated non-small-cell lung cancer. Lung Cancer. 2018 Jul;121:5-11. doi: 10.1016/j.lungcan.2018.04.012. Epub 2018 Apr 17. PMID 29858027